CLINICAL TRIAL: NCT00522925
Title: Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Safety and Efficacy of a Novel Dual Angiotensin and Endothelin Receptor Antagonist (PS433540) in Subjects With Stage I and II Hypertension
Brief Title: A Trial to Evaluate the Safety and Efficacy of PS433540 to Treat Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCO-C-008
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Results first posted 2011-09-14 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Hypertension
Keywords: hypertension; high blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Matching Placebo
  Interventions: Drug: placebo
- 2 (Experimental)
  Interventions: Drug: PS433540
- 3 (Experimental)
  Interventions: Drug: PS433540

INTERVENTIONS:
Drug: PS433540 — 200mg capsule, once daily for 28 days
  Arms: 2
Drug: placebo — placebo capsule, once daily for 28 days
  Arms: 1
Drug: PS433540 — 500mg capsule, once daily for 28 days
  Arms: 3

SUMMARY:
The purpose of the study is to see if PS433540 lowers blood pressure better than placebo and to see how safe PS433540 is compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 30 - 80 years
* Mean seated Systolic Blood Pressure (SBP) ≥ 150 - ≤ 179 mmHg and mean seated DBP < 110 mmHg at two consecutive qualifying visits. The mean difference in SBP between the two consecutive qualifying visits must be ≤ 10 mmHg.
* Mean daytime (8AM - 4PM) ambulatory SBP must be between ≥ 140 - ≤ 179 mmHg and mean daytime (8AM - 4PM) Diastolic Blood Pressure (DBP) ≤ 110 mmHg
* Subjects must have a usual daytime schedule. Night shift workers are excluded from participation.
* Women of child-bearing potential (WOCBP) and male subjects must use two reliable forms of contraception if sexually active. Alternatively, female subjects must be postmenopausal (for at least 1 year)

Exclusion Criteria:

* Subjects with serious disorders which may limit the ability to evaluate the efficacy or safety of PS433540, including cardiovascular, renal (including the absence of one kidney), pulmonary, hepatic, gastrointestinal (including clinically significant malabsorption), endocrine/metabolic, hematologic/oncologic (including an active malignancy other than basal cell carcinoma), neurologic and psychiatric diseases.
* Subjects with a history of myocardial infarction, angina, coronary angioplasty, bypass surgery or New York Heart Association (NYHA) class II-IV heart failure within the last 6 months.
* Subjects with a history of cerebrovascular accident or transient ischemic attack within the last 1 year.
* Subjects with diabetes mellitus (type I and type II).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Neutel, MD, Principal Investigator — Integrium
Locations (15):
- United States (15):
  - Premiere Pharmaceutical Research, LLC, Tempe, Arizona
  - Clinical Trials Research, Lincoln, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - National Research Institute, Los Angeles, California
  - Sacramento Research Medical Group, Sacramento, California
  - Orange County Research Center, Tustin, California
  - Westlake Medical Center, Westlake Village, California
  - University Clinical Research Deland, LLC, DeLand, Florida
  - Alan Graff, MD PA, Fort Lauderdale, Florida
  - Cedar Crosse Research Center, Chicago, Illinois
  - Orland Primary Care Specialists, Orland Park, Illinois
  - MD Medical Research, Oxon Hill, Maryland
  - Lindner Clinical Trial Center, Cincinnati, Ohio
  - Punzi Medical Center, Carrolton, Texas
  - Gemini Scientific, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- 1- Placebo: Placebo
- 2- PS433540 200mg: 200mg daily for 4 weeks
- 3- PS433540 500mg: 500mg once daily for 4 weeks
Period: Overall Study
Arm/Group | 1- Placebo | 2- PS433540 200mg | 3- PS433540 500mg
Started | 36 | 39 | 38
Completed | 28 | 38 | 36
Not Completed | 8 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1- Placebo | 2- PS433540 200mg | 3- PS433540 500mg | Total
Number analyzed (Participants) | 36 | 39 | 38 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 27 | 31 | 88
  >=65 years | 6 | 12 | 7 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 58.4 (7.94) | 59.1 (8.72) | 56.8 (9.87) | 58.1 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 10 | 40
  Male | 24 | 21 | 28 | 73
Region of Enrollment [Number; unit: participants]
  United States | 36 | 39 | 38 | 113

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean 24-hour Ambulatory Systolic Blood Pressure
Time Frame: 4 weeks of treatment with PS43540
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | 1- Placebo | 2- PS433540 200mg | 3- PS433540 500mg
Number analyzed (Participants) | 36 | 39 | 38
mmHg | -0.3 [-4.8 to 4.2] | -11.9 [-15.3 to -8.6] | -15.3 [-18.8 to -11.8]

2. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory Diastolic Blood Pressure
Time Frame: 4 weeks of treatment with PS43540
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in Mean Seated Systolic and Diastolic Blood Pressure
Time Frame: 4 weeks of treatment with PS43540
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | 1- Placebo | 2- PS433540 200mg | 3- PS433540 500mg
Serious Adverse Events (participants affected / at risk) | 1/36 | 1/39 | 0/38
Other Adverse Events (participants affected / at risk) | 9/36 | 8/39 | 10/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1- Placebo (N=36) | 2- PS433540 200mg (N=39) | 3- PS433540 500mg (N=38)
Syncope (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Syncope and confusional state in placebo patient that led to withdrawal
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — Reported prior to subject randomization
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1- Placebo (N=36) | 2- PS433540 200mg (N=39) | 3- PS433540 500mg (N=38)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (6) | 2 (2) | 3 (4)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Blood Pressure Increase (Investigations) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Oedema Peripheral (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No